CLINICAL TRIAL: NCT01930162
Title: A Single-arm, Open-label Study to Evaluate the Safety and Tolerability of Infusing HSC835 in Patients With Hematological Malignancies Undergoing UCB Transplantation Using a Non-myeloablative Conditioning Regimen
Brief Title: Safety and Tolerability of HSC835 in Patients With Hematological Malignancies Undergoing Single Umbilical Cord Blood Transplant
Acronym: UCBT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHSC835X2202
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2017-08-10 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2017-08

CONDITIONS: Single Umbilical Cord Blood Transplantation; Non-myeloablative Conditioning; Acute Lymphocytic Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma; Multiple Myeloma; Chronic Lymphocytic Leukemia
Keywords: HSC835; single umbilical cord blood transplantation; non-myeloablative conditioning regimen; Umbilical cord blood; UCB transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HSC835 (Experimental): Patients with hematologic malignancies requiring UCB transplant with a NMA conditioning regimen.
  Interventions: Drug: HSC835

INTERVENTIONS:
Drug: HSC835 — HSC835 is a stem cell therapy product providing a source of Hematopoietic stem cell (HSC).

SUMMARY:
This study was designed to evaluate the safety and tolerability of HSC835 for clinical use as measured by the absence of graft failure at day 42 in excess of that currently observed with double umbilical cord blood (UCB) transplantation (DUCBT) with non-myeloablative (NMA) conditioning.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis that qualifies them for UCBT
* Adequate organ function
* Availability of eligible donor material

Exclusion Criteria:

* Pregnancy or breastfeeding women and women of child-bearing potential unless two acceptable forms of contraception are being used
* Human immunodeficiency virus (HIV) infection
* Active infection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2016-08-29 (Actual); Study Completion 2016-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=183

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled into the study until approximately nine (9) patients were evaluable for safety as measured by the absence of infusional toxicity and sustained engraftment at Day 100.
Period: Overall Study
Arm/Group | HSC835
Started | 9
Completed | 4
Not Completed | 5
Not completed — Abnormal test procedure result(s) | 4
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: The Safety analysis included all enrolled patients who were transplanted with HSC835 (any patient with a date for HSC835 transplant).
Arm/Group | HSC835
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Absence of Graft Failure at Day 42
Description: This endpoint was to study safety and tolerability of HSC835 as measured by the absence of graft failure at day 42 in excess of that currently observed with double umbilical cord blood (UCB) transplantation (DUCBT) with non-myeloablative (NMA) conditioning.
Time Frame: 42 days
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | HSC835
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: Incidence of Neutrophil Recovery Within 42 Days
Description: Engraftment is defined as the first of three consecutive days with ANC > 0.5 x 109/L.
Time Frame: 42 days
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | HSC835
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Incidence of Non-relapse Mortality (NRM) Within 100 Days and One Year
Description: NRM includes all patients who died from any other cause except relapse of the underlying disease during the study duration.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | HSC835
Number analyzed (Participants) | 9
Participants | 1

4. Secondary Outcome: Incidence of Overall Survival Within One Year
Description: Overall survival is the proportion of patients who were alive at the end of the one year study period.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | HSC835
Number analyzed (Participants) | 9
Participants | 5

5. Secondary Outcome: Incidence of Relapse-free Survival Within One Year
Description: Patients are considered to have achieved relapse-free survival if they had not experienced either relapse or death (of any cause) at the end of the study.
Time Frame: 1 year
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | HSC835
Number analyzed (Participants) | 9
Participants | 4

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All Adverse Events reported in this record are from date of First Patient First Treatment until Last Patient Last Visit.
Groups:
- Time Period From Transplant Until 48hrs After Transplant: Adverse events that occurred within the first 48 hours of transplant.
- Time Period From Day 3 up to End of Study: Adverse Events that occurred 48 hours post-transplant.
Arm/Group | Time Period From Transplant Until 48hrs After Transplant | Time Period From Day 3 up to End of Study
Serious Adverse Events (participants affected / at risk) | 0/9 | 9/9
Other Adverse Events (participants affected / at risk) | 8/9 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Time Period From Transplant Until 48hrs After Transplant (N=9) | Time Period From Day 3 up to End of Study (N=9)
Oesophageal achalasia (Gastrointestinal disorders) | 0 | 1
Acute graft versus host disease (Immune system disorders) | 0 | 6
Cellulitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 2
Cytomegalovirus viraemia (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 0 | 1
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Transplant failure (Injury, poisoning and procedural complications) | 0 | 1
Chronic lymphocytic leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Time Period From Transplant Until 48hrs After Transplant (N=9) | Time Period From Day 3 up to End of Study (N=9)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cytomegalovirus viraemia (Infections and infestations) | 0 | 3
Enterococcal bacteraemia (Infections and infestations) | 0 | 3
Epstein-Barr viraemia (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
Methylobacterium infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 3 | 1
Headache (Nervous system disorders) | 3 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 4 | 0
Hypotension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.